CLINICAL TRIAL: NCT02890342
Title: The Natural History, Physiology, Microbiome and Biochemistry Studies of Propionic Acidemia
Brief Title: Natural History, Physiology, Microbiome and Biochemistry Studies of Propionic Acidemia
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160156; 16-HG-0156
Record Dates: First submitted 2016-09-03; First posted 2016-09-07 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-09-11

CONDITIONS: Metabolic Disease; Propionic Acidemia; Organic Acidemia
Keywords: Organic Acidemia; Inborn Errors of Metabolism; Natural History
MeSH Terms: conditions — Metabolic Diseases; Propionic Acidemia; Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected Patients with Propionic Acidemia: Patients with Propionic Acidemia, standard adult, parental permission
- Healthy Volunteers: Healthy Volunteers, standard adult, parental permission
- Unaffected Family Members: Unaffected family members

SUMMARY:
Background:

People s bodies need to break down food into the chemicals. These chemicals are used for energy and growth. Some people cannot process all chemicals very well. Too much of some chemicals can cause diseases. One of these diseases is called propionic acidemia (PA). People with PA can have problems with growth, learning heart, abdomen, and other organs. Researchers want to better understand how these problems happen.

Objective:

To learn more about propionic acidemia and the genes that might contribute to it.

Eligibility:

People at least 2 years old with PA who can travel to the clinic

Some unaffected family members

Design:

Participants will have a 3 to 5-day hospital visit every year or every few years. Family members may have just 1 visit.

During the family member visit, they may have:

Medical history

Physical exam

Samples of blood and urine

Questions about diet and a food diary

Doctors and nurses may do additional studies:

Samples of saliva, skin and stool

Fluid from a gastronomy tube, if participants have one

Dental and eye evaluations

A kidney test - a small amount of dye will be injected and blood will be collected.

Consultations with specialists

A test of calories needed at rest. A clear plastic tent is placed over the participant to measure breathing.

Stable isotope study. Participants will take a nonradioactive substance then blow into a bag.

Photos taken of the face and body with underwear on

Ultrasound of the abdomen

Heart tests

Hand x-ray

Brain scan

Participants may have other tests if study doctors recommend them. They will get the results of standard medical tests and genetic tests.

DETAILED DESCRIPTION:
Propionic acidemia (PA) is one of the most common inborn errors of organic acid metabolism. Although this disorder is now routinely detected in the immediate neonatal period on the US newborn screen, clinical outcomes are poor despite timely and aggressive medical intervention. Worldwide, the incidence of PA varies widely. The estimated live-birth incidence of PA is 1:243,000 in the US, 1:166,000 in Italy and 1:250,000 in Germany. Affected patients are medically fragile and can suffer from complications such as failure to thrive, intellectual disability, basal ganglia strokes, seizures, cardiomyopathy, cardiac arrhythmias, pancreatitis, impaired gut motility, osteoporosis and hematological complications. The frequency of these complications in the US patients and their precipitants remain poorly understood. Furthermore, current treatment outcomes have continued to demonstrate substantial morbidity and mortality in the patient population. Specific treatments include dietary modification to reduce propiogenic precursor load, levocarnitine to facilitate excretion of propionate, and oral antibiotics to suppress propionogenic gut flora. More recently, solid organ transplantation (liver and/or kidney) has been used to treat PA patients experiencing frequent and severe episodes of metabolic instability. However, optimal transplant strategy and post-transplant management have not been delineated. Several survey-based and retrospective studies describing the natural history of propionic acidemia have been published in the last decade. While these publications added to our understanding of the clinical course of this disease, these studies have not systematically focused on the US population using prospective analysis and reflect largely European experience, where many developed countries do not routinely screen for PA using newborn screen. Thus, the benefits of newborn screening on the PA outcomes require further clarification.

Under proposed NIH protocol, we will prospectively evaluate patients with propionic acidemia with special emphasis on the US population. Typical inpatient admissions and outpatient evaluations will last up to 4-5 days and may involve blood drawing, urine collection, stool collections, genomic studies, ophthalmological examination, cardiology evaluation, radiological procedures, brain and cardiac MRI/MRS, dietary assessment and neurobehavioral evaluation. In some patient s skin biopsies will be pursued.

The study objectives will be to describe the natural history of propionic acidemia in the US patients by delineating the spectrum of phenotypes and querying for genotype, enzymology, microbiome, and phenotype correlations. The population will consist of patients previously evaluated at NIH, physician referrals, and families directed to the study from clinicaltrials.gov, Organic Acidemia Association and Propionic Acidemia Foundation. Patients will be evaluated at the NIH Clinical Center or via telehealth platforms supported by NIH. Outcome measures will largely be descriptive and encompass correlations between clinical, microbiological, biochemical and molecular parameters.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients 2 years of age or older, of any gender and ethnicity, with propionic acidemia are eligible to enroll in this protocol. Patients diagnosis will be confirmed based on biochemical and/or molecular and enzymatic testing. Participants of any gender and ethnicity over 1 month of age are eligible to enroll remotely for collection of outside records and natural history data. They will be eligible to enroll in the full study for in-person evaluation at 2 years of age.
* Unaffected family members over 1 month of age, of any ethnicity or race, may be included in the study as household controls for microbiome studies and/or for genetic analysis. Studies in unaffected family members may include collection of medical and family history; if necessary completion of physical examination; drawing of blood for research purposes include testing of DNA; collection of stool samples for microbiome studies; collection of dietary history using pen-and-paper or electronic food diary and questionnaires; collection of saliva for metabolite and DNA analysis. In some unaffected family members without a known familial cause of propionic acidemia, exome sequencing or genome sequencing could be performed. Unaffected family members will not receive direct benefit from taking part in the study.
* If a participant becomes pregnant while on study, the participant can remain on study. The only way to learn more about the critical biological differences in those who affected with propionic acidemia who are pregnant is to continue to follow pregnant women on study.

However, no tests or procedures that are greater then minimal risk will be performed. Affected subjects who are pregnant may undergo procedures as part of their clinical care, including blood draws, genetic studies, and consultations, according to the clinical judgement of the clinical team. However, pregnant participants will be excluded from procedures such as organ tissue collection, stable isotope studies, GFR testing, and brain or cardiac MRI until the pregnancy is concluded.

* Healthy volunteers may be eligible to participate in the study if they are between 12 - 40 years of age, must meet specific BMI criteria (similar to affected individuals studied).
* Patients with propionic acidemia over 1 month of age, of any gender and ethnicity, undergoing a transplantation surgery at Children s Hospital of Pittsburgh, are eligible to participate in the tissue collection arm of the study.

EXCLUSION CRITERIA:

* The PI/AI may decline to enroll a patient because of poor metabolic control, lack of a primary metabolic/genetics physician, and intercurrent infection are exclusion criteria for this protocol, the likelihood that an acutely ill or poorly controlled patient will enroll will be minimized.
* A subset of participants may be enrolled in the tissue collection part of the study only (i.e. if they are too sick to travel). We can may also arrange limited remote consultation with our research team and NIH consultants, the participants referring physician and the participant/their legal guardian through the telephone or an NIH supported telehealth platform for participants who are unable to safely travel to NIH. This would not replace a study visit but would be used when travel isn t possible due to extenuating circumstances (e.g. pandemic). Participants would be encouraged to follow-up for a more thorough in-person evaluation when they are able to travel to NIH.
* For the healthy volunteers, they will be excluded if they have halitosis, cavities, dental or gingival problems, respiratory diseases (for example, asthma or recent history of COVID19), use tobacco products (for example, cigarette smoking or chewing tobacco), or use electronic nicotine delivery systems (for example, use of e-cigarettes or vaping devices), as this may interfere with accurate measurement of their volatile organic compounds. NIH staff and their family members will be eligible to participate in the healthy volunteer portion of the study.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Propionic Acidemia
Sampling Method: Non-Probability Sample
Enrollment: 1045 (Estimated)
Dates: Start 2016-11-29 (Actual); Primary Completion 2036-08-31 (Estimated); Study Completion 2036-08-31 (Estimated)

PRIMARY OUTCOMES:
Natural history to asess long term complications of Propionic Acidemia | Ongoing
  assessing the long term complications of Propionic Acidemia during a week long evaluation with imaging, labs, and consultations.

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Venditti, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Study is observational natural history study that is ongoing with no defined endpoints

REFERENCES:
- [Derived] Shchelochkov OA, Davies H, Mohney RP, Hatch A, Birch O, Ferry S, Van Ryzin C, Hall C, McCoy S, Vockley J, Kuo MJM, Manoli I, Sloan JL, Venditti CP. Breath biopsy in inborn errors of metabolism: A proof-of-principle study in propionic acidemia. Mol Genet Metab. 2025 Mar;144(3):109005. doi: 10.1016/j.ymgme.2024.109005. Epub 2024 Dec 21. PMID 39787887
- [Derived] Shchelochkov OA, Manoli I, Juneau P, Sloan JL, Ferry S, Myles J, Schoenfeld M, Pass A, McCoy S, Van Ryzin C, Wenger O, Levin M, Zein W, Huryn L, Snow J, Chlebowski C, Thurm A, Kopp JB, Chen KY, Venditti CP. Severity modeling of propionic acidemia using clinical and laboratory biomarkers. Genet Med. 2021 Aug;23(8):1534-1542. doi: 10.1038/s41436-021-01173-2. Epub 2021 May 18. PMID 34007002
- [Derived] Shchelochkov OA, Manoli I, Sloan JL, Ferry S, Pass A, Van Ryzin C, Myles J, Schoenfeld M, McGuire P, Rosing DR, Levin MD, Kopp JB, Venditti CP. Chronic kidney disease in propionic acidemia. Genet Med. 2019 Dec;21(12):2830-2835. doi: 10.1038/s41436-019-0593-z. Epub 2019 Jun 28. PMID 31249402
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-HG-0156.html